CLINICAL TRIAL: NCT03895307
Title: Comparison of Kinesio Taping and Local Injection in Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Abdulhamid Han Training and Research Hospital, Istanbul, Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ademerbirol
Record Dates: First submitted 2019-03-28; First posted 2019-03-29 (Actual); Results first posted 2020-07-02 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-03

CONDITIONS: Chronic Low Back Pain
Keywords: chronic low back pain; kinesio taping; injection; local anesthetic
MeSH Terms: interventions — Athletic Tape; Anesthetics, Local

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- kinesio taping (Experimental): two 15 cm I type kinesio tape applied longitudinally
  Interventions: Other: kinesio tape
- sham kinesio taping (Placebo Comparator): two 15 cm I type kinesio tape applied longitudinally but without stretching
  Interventions: Other: kinesio tape
- local anesthetic (Experimental): 18-20 cc %0.5 lidocaine subcutaneous injection
  Interventions: Other: local anesthetic
- local serum physiologic (Placebo Comparator): 18-20 cc % 0.09 NaCl subcutaneous injection
  Interventions: Other: local serum physiologic

INTERVENTIONS:
Other: kinesio tape — two 15 cm I type kinesio tape applied longitudinally
  Arms: kinesio taping; sham kinesio taping
Other: local anesthetic — local anesthetic: 18-20 cc %0.5 lidocaine subcutaneous injection
  Arms: local anesthetic
Other: local serum physiologic — serum physiologic : 18-20 cc % 0.09 NaCl subcutaneous injection
  Arms: local serum physiologic

SUMMARY:
Low back pain can be seen in every period of life. More than 80 percent of the society complain of low back pain at any time of life. Although the frequency of applying to a health institution due to low back pain varies from one society to the other, it takes place in the first three places in each community. Low back pain should be differentiated as new (acute) and long-term (chronic). In the treatment of chronic low back pain, rest, education, pharmacological treatment, physical therapy, painful point injections, surgical interventions, kinesio taping can be applied. The most frequently used physical therapy modalities for treatment of chronic low back pain are superficial and deep heat modalities (hot pack, infrared, ultrasound, microwave diathermy radar) and analgesic effective electrotherapy (TENS, interferential flows) modalities. One of the most important treatments is exercise therapy. In cases where conventional treatment of chronic low back pain is insufficient, that is, the patient's pain is still ongoing and functional recovery is insufficient, some alternative methods are also applied. These treatments include ozone, prolotherapy injection applications, dry needling, acupuncture, phytotherapy, balneotherapy, kinesio taping and so on. The aim of this study is to compare the efficacy of painful point injection and kinesio taping treatments in lumbar region in patients with chronic low back pain.

DETAILED DESCRIPTION:
Approximately 84 volunteer patients will be included in the study, patients older than 18 years, under 75 years of age, with a minimum of 3 months of mechanical back pain, Visual Analog Scale score of at least 60 patients will be included. Who are older than 18 years of age, having mental problems, having peripheral problems affecting the central nervous system, having received physical therapy to the lumbar region in the last 3 months, having been applied to the lumbar region within the last 3 months, having a history of lumbar region surgery, having a history of patients with motor deficit in the extremity, needle phobia, lidocaine and / or kinesio tape allergy, patients with wound, infection, burn, allergic lesions in the application area will not be included.

Patients included in the study will be included in the first (first), second (second), third (third) or fourth (fourth) treatment group by random number generator method.

The first group will be given the hot package (20 minutes / day) + exercise + 1. 4. 7. 10. 13. 16. days.

The second group will be given a hot package (20 minutes / day) + exercise + 1. 4. 7. 10. 13. 16 days.

The third group hot package (20 minutes / day) + exercise + 1. 4. 7. 10. 13. 16. days, kinesio tape will be applied to the determined areas.

the fourth group hot package (20 minutes / day) + exercise + 1. 4. 7. 10. 13. 16. days sham tape application will be made in the regions determined. ****

* Patients in all groups will continue to use the hotpack and exercises until the 3rd month after the first day of their study. First session exercises with the same physiotherapist (stretching for back-waist, iliopsoas and hamstring muscles; exercise range of hip and waist; hip and waist isometric exercises). Each patient will do the exercises 20 minutes after the hot package application.

  * saline and local anesthetic injection points to be applied to the lumbar region:

    1. Future points on spinous projections from L1 to L5
    2. Lumbar region 2 from the middle point of the spinous output bilateral and 2 cm to 4 cm lateral points
    3. To each point of the iliac lobe of iliac crest will be injected subcutaneously with 0.5 ml 0.5% lidocaine-containing local anesthetic.
    4. 6 mm 30 gauge needle tip will be used for injection.
    5. For each patient who underwent subcutaneous local anesthetic, an average of 18-20 ml of 0.5% lidocaine-containing local anesthetic and 18-20 ml of 0.09% NaCl-containing isotonic saline will be used for each patient.
    6. These points are the points of quadle technique applied in neural therapy.

       * Kinesio taping will use 2 cut-to-length I-bands with a length of about 15 cm long for one patient. Space correction technique will be used for patients. The lumbar region of the patients will be glued vertically to the paravertebral muscles vertically 3-4 cm lateral to the spinous projections. As a starting point for patients, S1 will be adhered to the vertebra without tension, then the patient will be asked to come with maximum lumbar flexion posterior.

         * For a patient in the treatment of sham kinesio taping, 2 pieces of approximately 15 cm long ends will be used to cut the curved I bands. The lumbar region of the patients will be glued vertically to the paravertebral muscles vertically 3-4 cm lateral to the spinous projections. Patients in the upright posture, kinesio tape S1 applied from the vertebra without stretching will be glued upwards and taped upwards.

ELIGIBILITY:
Inclusion Criteria:

1. Under 18 years of age under 75 years
2. Chronic mechanic (decreased with resting and resting) for at least 3 months
3. Visual Analogue Scale score of at least 60-

Exclusion Criteria:

1. Having mental problems
2. Having the disease affecting the peripheral and central nervous system
3. Have received physical therapy in the lumbar region within the last 3 months
4. Injection into the lumbar region within the last 3 months
5. Having a history of waist region surgery
6. Low motor dysfunction in lower extremity in physical examination
7. Needle phobia
8. Is allergic to lidocaine
9. Kinesio tape allergy
10. Wound, infection, burn, allergic lesions in the application area

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ADEM ERBİROL, Study Director — sultan abdulhamid han
Locations (2):
- Turkey (Türkiye) (2):
  - Sultan 2.Abdülhamid Han Training and Research Hospital, Istanbul, Eyalet/Yerleşke
  - Sultan Abdülhamid Han Training and Research Hospital, Istanbul, Eyalet/Yerleşke

IPD SHARING:
Plan to Share IPD: No
other researchers would get information from the main researcher. therefore it was not shared.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Kinesio Taping | Sham Kinesio Taping | Local Anesthetic | Local Serum Physiologic
Started | 21 | 20 | 22 | 21
Completed | 19 | 20 | 20 | 21
Not Completed | 2 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Kinesio Taping | Sham Kinesio Taping | Local Anesthetic | Local Serum Physiologic | Total
Number analyzed (Participants) | 21 | 20 | 22 | 21 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 17 | 17 | 20 | 74
  >=65 years | 1 | 3 | 5 | 1 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.67 (15.72) | 47.20 (16.60) | 47.82 (15.95) | 41.48 (15.69) | 44.05 (16.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 5 | 12 | 34
  Male | 12 | 12 | 17 | 9 | 50
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 21 | 20 | 22 | 21 | 84
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Turkey | 21 | 20 | 22 | 21 | 84
Body Mass Index [Mean (Standard Deviation); unit: kg/m2] | 27.63 (4.70) | 27.25 (3.88) | 27.05 (4.47) | 27.05 (3.73) | 27.24 (4.13)

OUTCOME MEASURES:

1. Primary Outcome: Pain Severity: Visual Analog Scale
Description: visual analog scale: minimum score: 0 maximum score: 10. Higher scores reflect more severe pain
Time Frame: day 0 (before intervention)
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Kinesio Taping | Sham Kinesio Taping | Local Anesthetic | Local Serum Physiologic
Number analyzed (Participants) | 21 | 20 | 22 | 21
score on a scale | 7.26 (0.8) | 7.75 (0.44) | 7.8 (0.89) | 7.62 (0.92)

2. Primary Outcome: Pain Severity: Visual Analog Scale
Description: visual analog scale: minimum score: 0 maximum score: 10. Higher scores reflect more severe pain
Time Frame: day 16 (after 6th application)
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Kinesio Taping | Sham Kinesio Taping | Local Anesthetic | Local Serum Physiologic
Number analyzed (Participants) | 19 | 20 | 20 | 21
score on a scale | 2.89 (2.1) | 3.35 (2.11) | 2.85 (1.98) | 3.52 (2.13)

3. Primary Outcome: Pain Severity: Visual Analog Scale
Description: visual analog scale: minimum score: 0 maximum score: 10. Higher scores reflect more severe pain
Time Frame: 1 month after intervention
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Kinesio Taping | Sham Kinesio Taping | Local Anesthetic | Local Serum Physiologic
Number analyzed (Participants) | 19 | 20 | 20 | 21
score on a scale | 3.58 (2.56) | 4.65 (2.99) | 3.65 (2.36) | 5.81 (2.18)

4. Primary Outcome: Pain Severity: Visual Analog Scale
Description: visual analog scale: minimum score: 0 maximum score: 10. Higher scores reflect more severe pain
Time Frame: 3 months after intervention
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Kinesio Taping | Sham Kinesio Taping | Local Anesthetic | Local Serum Physiologic
Number analyzed (Participants) | 19 | 20 | 20 | 21
score on a scale | 4.42 (2.41) | 5.20 (2.94) | 5 (2.77) | 6.48 (2.22)

5. Secondary Outcome: Disability Severity: Oswestry Disabiliy Index
Description: Oswestry Disabiliy Index:
  minimum score: 0 maximum score: 50. Higher scores reflect more severe disability
Time Frame: day 0 (before intervention)
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Kinesio Taping | Sham Kinesio Taping | Local Anesthetic | Local Serum Physiologic
Number analyzed (Participants) | 21 | 20 | 22 | 21
score on a scale | 17.42 (2.65) | 18.30 (3.45) | 17.1 (2.38) | 17.57 (1.72)

6. Secondary Outcome: Disability Severity: Oswestry Disability Index
Description: Oswestry Disabiliy Index:
  minimum score: 0 maximum score: 50. Higher scores reflect more severe disability
Time Frame: day 16 (after 6th application)
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Kinesio Taping | Sham Kinesio Taping | Local Anesthetic | Local Serum Physiologic
Number analyzed (Participants) | 19 | 20 | 20 | 21
score on a scale | 7.68 (6.67) | 6.50 (6.66) | 6.15 (4.95) | 10.43 (5.07)

7. Secondary Outcome: Disability Severity: Oswestry Disability Index
Description: Oswestry Disabiliy Index:
  minimum score: 0 maximum score: 50. Higher scores reflect more severe disability
Time Frame: 1 month after intervention
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Kinesio Taping | Sham Kinesio Taping | Local Anesthetic | Local Serum Physiologic
Number analyzed (Participants) | 19 | 20 | 20 | 21
score on a scale | 10.84 (8.21) | 10.50 (7.58) | 8.85 (6.67) | 14.38 (4.57)

8. Secondary Outcome: Disability Severity: Oswestry Disability Index
Description: Oswestry Disabiliy Index:
  minimum score: 0 maximum score: 50. Higher scores reflect more severe disability
Time Frame: 3 months after intervention
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Kinesio Taping | Sham Kinesio Taping | Local Anesthetic | Local Serum Physiologic
Number analyzed (Participants) | 19 | 20 | 20 | 21
score on a scale | 13.84 (6.44) | 14.20 (6.52) | 13.35 (4.35) | 16.10 (3.89)

9. Secondary Outcome: Patient Reported Quality of Life: Short Form 36 Physical Functioning
Description: short form 36: The SF-36 form generates eight subscales. The eight subscales are: physical functioning, role limitations due to physical problems, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health.
  short form 36 physical functioning subscale scores are given. minimum score: 0 maximum score: 100. Higher scores indicate a better of quality of life
Time Frame: day 0 (before intervention)
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Kinesio Taping | Sham Kinesio Taping | Local Anesthetic | Local Serum Physiologic
Number analyzed (Participants) | 21 | 20 | 22 | 21
score on a scale | 53.1 (13.08) | 50.75 (14.53) | 45.9 (12.54) | 50.71 (12.97)

10. Secondary Outcome: Patient Reported Quality of Life: Short Form 36 Physical Functioning
Description: as for outcome 9
Time Frame: day 16 (after 6th application)
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Kinesio Taping | Sham Kinesio Taping | Local Anesthetic | Local Serum Physiologic
Number analyzed (Participants) | 19 | 20 | 20 | 21
score on a scale | 77.63 (14.75) | 74 (13.53) | 75 (15.39) | 74.05 (15.46)

11. Secondary Outcome: Patient Reported Quality of Life: Short Form 36 Physical Functioning
Description: as for outcome 9
Time Frame: 1 month after intervention
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Kinesio Taping | Sham Kinesio Taping | Local Anesthetic | Local Serum Physiologic
Number analyzed (Participants) | 19 | 20 | 20 | 21
score on a scale | 68.11 (16.69) | 61.70 (19.47) | 67.20 (16.26) | 57.86 (16.32)

12. Secondary Outcome: Patient Reported Quality of Life: Short Form 36 Physical Functioning
Description: as for outcome 9
Time Frame: 3 months after intervention
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Kinesio Taping | Sham Kinesio Taping | Local Anesthetic | Local Serum Physiologic
Number analyzed (Participants) | 19 | 20 | 20 | 21
score on a scale | 58.84 (13.26) | 55.15 (15.35) | 56.65 (16.27) | 54.05 (14.63)

13. Secondary Outcome: Spinal Mobility: Schober Test
Description: Schober's test is classically used to determine if there is a decrease in lumbar spine range of motion (flexion).
  Patient is standing, examiner marks the L5 spinous process by drawing a horizontal line across the patients back.
  A second line is marked 10 cm above the first line. Patient is then instructed to flex forward as if attempting to touch his/her toes, examiner remeasures distance between two lines with patient fully flexed.
  The difference between the measurements in erect and flexion positions indicates the outcome of the lumbar flexion.
  Less than 5cm increase in length with forward flexion: Decreased lumbar spine range of motion.
Time Frame: day 0 (before intervention)
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Kinesio Taping | Sham Kinesio Taping | Local Anesthetic | Local Serum Physiologic
Number analyzed (Participants) | 21 | 20 | 22 | 21
centimeters | 4.09 (0.58) | 4.37 (0.77) | 3.75 (0.88) | 4.38 (0.72)

14. Secondary Outcome: Spinal Mobility: Schober Test
Description: as for outcome 13
Time Frame: day 16 (after 6th application)
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Kinesio Taping | Sham Kinesio Taping | Local Anesthetic | Local Serum Physiologic
Number analyzed (Participants) | 19 | 20 | 20 | 21
centimeters | 4.36 (0.43) | 4.37 (0.77) | 4.27 (0.63) | 4.59 (0.49)

15. Secondary Outcome: Spinal Mobility: Schober Test
Description: as for outcome 13
Time Frame: 1 month after intervention
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Kinesio Taping | Sham Kinesio Taping | Local Anesthetic | Local Serum Physiologic
Number analyzed (Participants) | 19 | 20 | 20 | 21
centimeters | 4.36 (0.43) | 4.42 (0.74) | 4.27 (0.63) | 4.54 (0.54)

16. Secondary Outcome: Spinal Mobility: Schober Test
Description: as for outcome 13
Time Frame: 3 months after intervention
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Kinesio Taping | Sham Kinesio Taping | Local Anesthetic | Local Serum Physiologic
Number analyzed (Participants) | 19 | 20 | 20 | 21
centimeters | 4.36 (0.43) | 4.42 (0.74) | 4.2 (0.61) | 4.54 (0.54)

17. Secondary Outcome: Patient Reported Quality of Life: Short Form-36 Mental Health
Description: Short Form 36: The SF-36 form generates eight subscales. The eight subscales are: physical functioning, role limitations due to physical problems, bodily pain, general health perceptions, vitality, social functioning, role limitations due to emotional problems, and mental health.
  Short Form-36 Mental health subscale scores are given. Mental minimum score: 0 maximum score: 100. Higher scores indicate a better of quality of life.
Time Frame: day 0 before intervention
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Kinesio Taping | Sham Kinesio Taping | Local Anesthetic | Local Serum Physiologic
Number analyzed (Participants) | 21 | 20 | 22 | 21
score on a scale | 68 (0) | 67.5 (2.23) | 68 (0) | 68 (0)

18. Secondary Outcome: Patient Reported Quality of Life: Short Form-36 Mental Health
Description: as for outcome 17
Time Frame: day 16 (after 6th application)
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Kinesio Taping | Sham Kinesio Taping | Local Anesthetic | Local Serum Physiologic
Number analyzed (Participants) | 19 | 20 | 20 | 21
score on a scale | 79.79 (7.48) | 78.6 (5.51) | 78 (5.51) | 77.52 (2.18)

19. Secondary Outcome: Patient Reported Quality of Life: Short Form-36 Mental Health
Description: as for outcome 17
Time Frame: 1 month after intervention
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Kinesio Taping | Sham Kinesio Taping | Local Anesthetic | Local Serum Physiologic
Number analyzed (Participants) | 19 | 20 | 20 | 21
score on a scale | 77.16 (9.29) | 73.10 (7.96) | 76.6 (7.05) | 71.81 (4.97)

20. Secondary Outcome: Patient Reported Quality of Life: Short Form-36 Mental Health
Description: as for outcome 17
Time Frame: 3 months after intervention
Population: intent to treat population(all participants)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Kinesio Taping | Sham Kinesio Taping | Local Anesthetic | Local Serum Physiologic
Number analyzed (Participants) | 19 | 20 | 20 | 21
score on a scale | 74.42 (7.96) | 72.1 (7.90) | 73.60 (7.93) | 71.33 (4.83)

ADVERSE EVENTS:
Time Frame: adverse events were not monitored/assessed
Description: adverse events were not monitored/assessed
Arm/Group | Kinesio Tape | Sham Kinesio Taping | Local Anesthetic | Local Serum Physiologic
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT03895307/Prot_SAP_000.pdf